CLINICAL TRIAL: NCT04341584
Title: CORIMUNO-ANA: Trial Evaluating Efficacy Of Anakinra In Patients With Covid-19 Infection, Nested In The CORIMUNO-19
Brief Title: CORIMUNO-ANA: Trial Evaluating Efficacy Of Anakinra In Patients With Covid-19 Infection
Acronym: CORIMUNO-ANA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP200375-5
Record Dates: First submitted 2020-04-07; First posted 2020-04-10 (Actual); Results first posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2020-04

CONDITIONS: Corona Virus Infection
MeSH Terms: conditions — Coronavirus Infections | interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ANAKINRA -- Severe COVID Population (WHO-Clinical Progression Scale =5 at baseline) (Experimental): Treatment includes the administration of Two IV infusions / day of ANAKINRA KINERET® 200mg (Total 400 mg) at day 1 (D1), D2 and D3, two IV infusions / day of ANAKINRA KINERET® 100mg (Total 200 mg) at day 4 (D4), and one IV infusion of ANAKINRA KINERET® 100mg (Total 100 mg) at day 5 (D5).
  In case of absence of improvement at D4 (absence of clinical improvement AND absence of decrease of CRP level > 50%), 3 supplementary days of treatment at 400 mg/day will be done at D4, D5, D6 followed by a decrease at 200 mg/day at D7 and 100 mg/day at D8 and stop thereafter
  Interventions: Drug: Anakinra
- Standard of care -- Severe COVID Population (WHO-Clinical Progression Scale =5 at baseline) (No Intervention)
- ANAKINRA -- Critical COVID Population (WHO-Clinical Progression Scale >5 at baseline) (Experimental): Treatment includes the administration of Two IV infusions / day of ANAKINRA KINERET® 200mg (Total 400 mg) at day 1 (D1), D2 and D3, two IV infusions / day of ANAKINRA KINERET® 100mg (Total 200 mg) at day 4 (D4), and one IV infusion of ANAKINRA KINERET® 100mg (Total 100 mg) at day 5 (D5).
  In case of absence of improvement at D4 (absence of clinical improvement AND absence of decrease of CRP level > 50%), 3 supplementary days of treatment at 400 mg/day will be done at D4, D5, D6 followed by a decrease at 200 mg/day at D7 and 100 mg/day at D8 and stop thereafter
  Interventions: Drug: Anakinra
- Standard of care -- Critical COVID Population (WHO-Clinical Progression Scale >5 at baseline) (No Intervention)

INTERVENTIONS:
Drug: Anakinra — Treatment includes the administration of Two IV infusions / day of ANAKINRA KINERET® 200mg (Total 400 mg) at day 1 (D1), D2 and D3, two IV infusions / day of ANAKINRA KINERET® 100mg (Total 200 mg) at day 4 (D4), and one IV infusion of ANAKINRA KINERET® 100mg (Total 100 mg) at day 5 (D5).
  In case of absence of improvement at D4 (absence of clinical improvement AND absence of decrease of CRP level > 50%), 3 supplementary days of treatment at 400 mg/day will be done at D4, D5, D6 followed by a decrease at 200 mg/day at D7 and 100 mg/day at D8 and stop thereafter
  Arms: ANAKINRA -- Critical COVID Population (WHO-Clinical Progression Scale >5 at baseline); ANAKINRA -- Severe COVID Population (WHO-Clinical Progression Scale =5 at baseline)

SUMMARY:
The overall objective of the study is to determine the therapeutic effect and tolerance of Anakinra in patients with moderate, severe pneumonia or critical pneumonia associated with Coronavirus disease 2019 (COVID-19). Anakinra (ANA) is a recombinant human decoy IL-1Ra and therefore blocks IL-1α and IL-1β. The study has a cohort multiple Randomized Controlled Trials (cmRCT) design. Randomization will occur prior to offering Anakinra administration to patients enrolled in the CORIMUNO-19 cohort. Anakinra will be administered to consenting adult patients hospitalized with CORVID-19 either diagnosed with moderate or severe pneumonia requiring no mechanical ventilation or critical pneumonia requiring mechanical ventilation. Patients who will chose not to receive Anakinra will receive standard of cares. Outcomes of Anakinra -treated patients will be compared with outcomes of standard of care treated patients as well as outcomes of patients treated with other immune modulators.

ELIGIBILITY:
Inclusion Criteria:

1. Patients included in the CORIMUNO-19 cohort
2. Patients with C-reactive protein level (CRP) > 25 mg / L the day or the day before the infusion)
3. Patients belonging to one of the 2 following groups:

   * Group 1: patients meeting all of the following criteria: 1) Requiring more than 3L/min of oxygen; 2) WHO progression scale = 5; 3) No non invasive ventilation or High flow
   * Group 2: patients with respiratory failure AND (requiring mechanical ventilation OR non invasive ventilation OR High flow), with a WHO progression scale ≥ 6, and no do-not-resuscitate (DNR) order

Exclusion Criteria:

* Patients with exclusion criteria to the CORIMUNO-19 cohort.
* Known hypersensitivity to Anakinra or to any of their excipients.
* Pregnancy
* Current documented bacterial infection.
* Patient with any of following laboratory results out of the ranges detailed below at screening:

  * Absolute neutrophil count (ANC) ≤ 1.0 x 109/L
  * Haemoglobin level: no limitation
  * Platelets (PLT) < 50 G /L
  * SGOT or SGPT > 5N
  * Severe renal insufficiency with Glomerular filtration rate < 30 ml / mn

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2020-04-08 (Actual); Primary Completion 2020-05-10 (Actual); Study Completion 2020-07-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Mariette, MD, PhD, Principal Investigator — Hôpital Bicêtre, Assistance Publique-Hôpitaux de Paris
Locations (1):
- Hôpital Bicêtre, Assistance Publique-Hôpitaux de Paris, Le Kremlin-Bicêtre, France

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] CORIMUNO-19 Collaborative group. Effect of anakinra versus usual care in adults in hospital with COVID-19 and mild-to-moderate pneumonia (CORIMUNO-ANA-1): a randomised controlled trial. Lancet Respir Med. 2021 Mar;9(3):295-304. doi: 10.1016/S2213-2600(20)30556-7. Epub 2021 Jan 22. PMID 33493450
- [Derived] Joly C, Desjardins D, Porcher R, Pere H, Bruneau T, Zhang Q, Bastard P, Cobat A, Resmini L, Lenoir O, Savale L, Lecuroux C, Verstuyft C, Roque-Afonso AM, Veyer D, Baron G, Resche-Rigon M, Ravaud P, Casanova JL, Le Grand R, Hermine O, Tharaux PL, Mariette X. More rapid blood interferon alpha2 decline in fatal versus surviving COVID-19 patients. Front Immunol. 2023 Nov 21;14:1250214. doi: 10.3389/fimmu.2023.1250214. eCollection 2023. PMID 38077399

RESULTS

PARTICIPANT FLOW:
Groups:
- ANAKINRA -- Severe COVID Population (WHO-CPS =5); ANAKINRA -- Critical COVID Population (WHO-CPS >5): Treatment includes the administration of Two IV infusions / day of ANAKINRA KINERET® 200mg (Total 400 mg) at day 1 (D1), D2 and D3, two IV infusions / day of ANAKINRA KINERET® 100mg (Total 200 mg) at day 4 (D4), and one IV infusion of ANAKINRA KINERET® 100mg (Total 100 mg) at day 5 (D5).
  In case of absence of improvement at D4 (absence of clinical improvement AND absence of decrease of CRP level > 50%), 3 supplementary days of treatment at 400 mg/day will be done at D4, D5, D6 followed by a decrease at 200 mg/day at D7 and 100 mg/day at D8 and stop thereafter
  Anakinra: Treatment includes the administration of Two IV infusions / day of ANAKINRA KINERET® 200mg (Total 400 mg) at day 1 (D1), D2 and D3, two IV infusions / day of ANAKINRA KINERET® 100mg (Total 200 mg) at day 4 (D4), and one IV infusion of ANAKINRA KINERET® 100mg (Total 100 mg) at day 5 (D5).
  In case of absence of improvement at D4 (absence of clinical improvement AND absence of decrease of CRP level > 50%), 3 supplementary days of treatment at 400 mg/day will be done at D4, D5, D6 followed by a decrease at 200 mg/day at D7 and 100 mg/day at D8 and stop thereafter
- Standard of Care -- Severe COVID Population (WHO-CPS =5); Standard of Care -- Critical COVID Population (WHO-CPS >5): Usual care was provided at the discretion of the site clinicians
Period: Overall Study
Arm/Group | ANAKINRA -- Severe COVID Population (WHO-CPS =5) | Standard of Care -- Severe COVID Population (WHO-CPS =5) | ANAKINRA -- Critical COVID Population (WHO-CPS >5) | Standard of Care -- Critical COVID Population (WHO-CPS >5)
Started | 59 | 57 | 24 | 21
Completed | 59 | 55 | 22 | 20
Not Completed | 0 | 2 | 2 | 1
Not completed — Withdrew consent | 0 | 2 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ANAKINRA -- Severe COVID Population (WHO-CPS =5) | Standard of Care -- Severe COVID Population (WHO-CPS =5) | ANAKINRA -- Critical COVID Population (WHO-CPS >5) | Standard of Care -- Critical COVID Population (WHO-CPS >5) | Total
Number analyzed (Participants) | 59 | 55 | 22 | 20 | 156
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 67 [55.5 to 74.3] | 64.9 [59.5 to 78.3] | 59.6 [54.4 to 68.5] | 61.5 [53.9 to 70] | 64.7 [57 to 73.2]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 18 | 7 | 5 | 46
  Male | 43 | 37 | 15 | 15 | 110
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body Mass Index >= 30 kg/m² [Count of Participants; unit: Participants] — Population: Missing data are possible
  Participants
    number analyzed (Participants) | 58 | 55 | 22 | 20 | 155
    (all) | 13 | 15 | 7 | 8 | 43
Weight [Median (Inter-Quartile Range); unit: kg] — Population: Missing data are possible
  kg
    number analyzed (Participants) | 59 | 46 | 22 | 20 | 147
    (all) | 78 [67 to 91] | 77.5 [70 to 95] | 81 [75 to 91] | 85 [80 to 91] | 80 [70 to 91]
SPO2 [Median (Inter-Quartile Range); unit: %] | 95 [93 to 97] | 95 [93 to 97] | 94.5 [92 to 98] | 94.5 [92 to 97] | 95 [93 to 97]
Temperature [Median (Inter-Quartile Range); unit: °C] | 37.8 [36.7 to 38.8] | 37.6 [37 to 38.5] | 37.8 [37 to 38.9] | 38.3 [37.4 to 39] | 37.8 [37 to 38.7]
Respiratory rate [Median (Inter-Quartile Range); unit: breaths/min] — Population: Missing data are possible
  breaths/min
    number analyzed (Participants) | 55 | 50 | 22 | 19 | 146
    (all) | 28 [24 to 32] | 28 [23 to 36] | 30 [25 to 35] | 26 [26 to 32] | 28 [24 to 32]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Non-invasive Ventilation, Mechanical Ventilation or Death at Day 14 -- Severe COVID Population (WHO Clinical Progression Scale =5 at Baseline)
Description: Survival without needs of ventilator utilization (including non invasive ventilation and high flow) at day 14. Percentage of non-invasive ventilation, mechanical ventilation or death. Thus, events considered are needing ventilator utilization (mechanical or non-invasive ventilation including high flow oxygen), or death. New do-not-resuscitate (DNR) order (if given after the inclusion of the patient) will be considered as an event at the date of the DNR.
Time Frame: Day 1 to Day 14
Population: Severe COVID population ((WHO clinical progression scale =5 at baseline)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ANAKINRA -- Severe COVID Population (WHO-CPS =5) | Standard of Care -- Severe COVID Population (WHO-CPS =5)
Number analyzed (Participants) | 59 | 55
percentage of participants | 47 [33 to 59] | 51 [36 to 62]
Statistical Analysis 1: Comparison: ANAKINRA -- Severe COVID Population (WHO-CPS =5) vs Standard of Care -- Severe COVID Population (WHO-CPS =5); Test type: Superiority; Bayesian Cox model; adjusted for age and centre; Median posterior HR = 0.97, 90% CI 2-sided [0.62 to 1.52] — % Confidence Interval is % Credible Interval here

2. Primary Outcome: Percentage of Participants With WHO Clinical Progression Scale > 5 at Day 4 -- Severe COVID Population (WHO Clinical Progression Scale =5 at Baseline)
Description: Percentage of participants who has died or needed non-invasive or mechanical ventilation by day 4 (WHO clinical progression scale > 5). A patient with new do-not-resuscitate order at day 4 will be considered as with a score > 5.
Time Frame: 4 days
Population: Severe COVID population (WHO clinical progression scale =5 at baseline)
Measure: Number; unit: percentage of participants
Arm/Group | ANAKINRA -- Severe COVID Population (WHO-CPS =5) | Standard of Care -- Severe COVID Population (WHO-CPS =5)
Number analyzed (Participants) | 59 | 55
percentage of participants | 36 | 38
Statistical Analysis 1: Comparison: ANAKINRA -- Severe COVID Population (WHO-CPS =5) vs Standard of Care -- Severe COVID Population (WHO-CPS =5); Test type: Superiority; Bayesian analysis; Median posterior absolute risk differenc = -2.5, 90% CI 2-sided [-17.1 to 12] — % Confidence Interval is % Credible Interval here

3. Primary Outcome: Cumulative Incidence (Percentage) of Participants With Successful Tracheal Extubation at Day 14 -- Critical COVID Population (WHO Clinical Progression Scale >5 at Baseline)
Description: Cumulative incidence (percentage) of successful tracheal extubation (defined as duration extubation > 48h) at day 14 if patients have been intubated before day 14 ; or removal of non invasive ventilation or high flow (for > 48h) if they were included under oxygen by non invasive ventilation or High flow (score 6) and remained without intubation. Death or new do-not-resuscitate order (if given after the inclusion of the patient) will be considered as a competing event.
Time Frame: Day 1 to Day 14
Population: Critical COVID population (WHO clinical progression scale >5 at baseline)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ANAKINRA -- Critical COVID Population (WHO-CPS >5) | Standard of Care -- Critical COVID Population (WHO-CPS >5)
Number analyzed (Participants) | 22 | 20
percentage of participants | 50 [28 to 69] | 40 [19 to 61]
Statistical Analysis 1: Comparison: ANAKINRA -- Critical COVID Population (WHO-CPS >5) vs Standard of Care -- Critical COVID Population (WHO-CPS >5); Test type: Superiority; Bayesian Fine and Gray analysis — adjusted for age and centre; Median posterior HR = 1.26, 90% CI 2-sided [0.59 to 2.81] — % Confidence interval is % Credible Interval here

4. Primary Outcome: Percentage of Participants With a Decrease of at Least One Point in WHO Clinical Progression Scale Score at Day 4 -- Critical COVID Population (WHO Clinical Progression Scale >5)
Description: Percentage of patients with a decrease of WHO score of at least 1 point at day 4
Time Frame: 4 days
Population: Critical COVID population (WHO clinical progression scale >5)
Measure: Number; unit: percentage of participants
Arm/Group | ANAKINRA -- Critical COVID Population (WHO-CPS >5) | Standard of Care -- Critical COVID Population (WHO-CPS >5)
Number analyzed (Participants) | 22 | 20
percentage of participants | 36 | 10
Statistical Analysis 1: Comparison: ANAKINRA -- Critical COVID Population (WHO-CPS >5) vs Standard of Care -- Critical COVID Population (WHO-CPS >5); Test type: Superiority; Bayesian analysis; Median posterior absolute risk differenc = 24, 90% CI 2-sided [3.9 to 43.5] — % Confidence interval is % Credible interval here

5. Secondary Outcome: WHO Clinical Progression Scale
Description: WHO clinical progression scale: Uninfected; non viral RNA detected: 0 Asymptomatic; viral RNA detected: 1 Symptomatic; Independent: 2 Symptomatic; Assistance needed: 3 Hospitalized; No oxygen therapy: 4 Hospitalized; oxygen by mask or nasal prongs: 5 Hospitalized; oxygen by Non invasive Ventilation or High flow: 6 Intubation and Mechanical ventilation, pO2/FIO2>=150 OR SpO2/FIO2>=200: 7 Mechanical ventilation, (pO2/FIO2<150 OR SpO2/FIO2<200) OR vasopressors (norepinephrine >0.3 microg/kg/min): 8 Mechanical ventilation, pO2/FIO2<150 AND vasopressors (norepinephrine >0.3 microg/kg/min), OR Dialysis OR ECMO: 9 Dead: 10.
Time Frame: 4, 7, 14, 28 days
Population: No comparison was planned at Day 7 in the Severe COVID Population (WHO clinical progression scale =5) so no descriptive/comparative data were done. No comparison was planned at Day 28 in Critical COVID Population (WHO clinical progression scale >5) so no descriptive/comparative data were done.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | ANAKINRA -- Severe COVID Population (WHO-CPS =5) | Standard of Care -- Severe COVID Population (WHO-CPS =5) | ANAKINRA -- Critical COVID Population (WHO-CPS >5) | Standard of Care -- Critical COVID Population (WHO-CPS >5)
Number analyzed (Participants) | 59 | 55 | 22 | 20
units on a scale
  Day 4 | 5 [5 to 6] | 5 [5 to 6] | 7 [6 to 8] | 6 [6 to 8]
  Day 7 | NA [NA to NA] — No comparison was planned at Day 7 in the Severe COVID Population (WHO clinical progression scale =5) so no descriptive/comparative data were done. | NA [NA to NA] — No comparison was planned at Day 7 in the Severe COVID Population (WHO clinical progression scale =5) so no descriptive/comparative data were done. | 7 [6 to 8] | 7 [5 to 8]
  Day 14: number analyzed (Participants) | 54 | 53 | 22 | 20
  Day 14 | 5 [5 to 7] | 5 [5 to 7] | 6 [4 to 8] | 6 [5 to 8]
  Day 28: number analyzed (Participants) | 56 | 53 | 22 | 20
  Day 28 | 5 [2 to 8] | 5 [3 to 8] | NA [NA to NA] — No comparison was planned at Day 28 in Critical COVID Population (WHO clinical progression scale >5) so no descriptive/comparative data were done. | NA [NA to NA] — No comparison was planned at Day 28 in Critical COVID Population (WHO clinical progression scale >5) so no descriptive/comparative data were done.
Statistical Analysis 1: Comparison: ANAKINRA -- Severe COVID Population (WHO-CPS =5) vs Standard of Care -- Severe COVID Population (WHO-CPS =5); Day 4; Test type: Superiority; Bayesian Proportionnal odds model; Adjusted for age and centre; Median posterior OR = 0.80, 95% CI 2-sided [0.38 to 1.68] — % Confidence interval is % Credible interval here
Statistical Analysis 2: Comparison: ANAKINRA -- Severe COVID Population (WHO-CPS =5) vs Standard of Care -- Severe COVID Population (WHO-CPS =5); Day 14; Test type: Superiority; Bayesian Proportionnal odds model; Adjusted for age and centre; Median posterior OR = 0.69, 95% CI 2-sided [0.33 to 1.43] — % Confidence interval is % Credible interval here
Statistical Analysis 3: Comparison: ANAKINRA -- Severe COVID Population (WHO-CPS =5) vs Standard of Care -- Severe COVID Population (WHO-CPS =5); Day 28; Test type: Superiority; Bayesian Proportionnal odds model; Adjusted for age and centre; Median posterior OR = 0.70, 95% CI 2-sided [0.35 to 1.38] — % Confidence interval is % Credible interval here
Statistical Analysis 4: Comparison: ANAKINRA -- Critical COVID Population (WHO-CPS >5) vs Standard of Care -- Critical COVID Population (WHO-CPS >5); Day 4; Test type: Superiority; Bayesian Proportionnal odds model; Adjusted for age and centre; Median posterior OR = 0.72, 95% CI 2-sided [0.22 to 2.39] — % Confidence Interval is % Credible interval here
Statistical Analysis 5: Comparison: ANAKINRA -- Critical COVID Population (WHO-CPS >5) vs Standard of Care -- Critical COVID Population (WHO-CPS >5); Day 7; Test type: Superiority; Bayesian Proportionnal odds model; Adjusted for age and centre; Median posterior HR = 0.89, 95% CI 2-sided [0.28 to 2.80] — % Confidence Interval is % Credible interval here
Statistical Analysis 6: Comparison: ANAKINRA -- Critical COVID Population (WHO-CPS >5) vs Standard of Care -- Critical COVID Population (WHO-CPS >5); Test type: Superiority; Bayesian Proportionnal odds model — Day 14; Adjusted for afe and centre; Median posterior HR = 0.57, 95% CI 2-sided [0.18 to 1.75] — % Confidence Interval is % Credible interval here

6. Secondary Outcome: Percentage of Participants Surviving (Overall Survival)
Description: Percentage of participants surviving at 14, 28 and 90 days
Time Frame: 14, 28 and 90 days
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- ANAKINRA -- Critical COVID Population (WHO-CPS >5): Treatment includes the administration of Two IV infusions / day of ANAKINRA KINERET® 200mg (Total 400 mg) at day 1 (D1), D2 and D3, two IV infusions / day of ANAKINRA KINERET® 100mg (Total 200 mg) at day 4 (D4), and one IV infusion of ANAKINRA KINERET® 100mg (Total 100 mg) at day 5 (D5).
  In case of absence of improvement at D4 (absence of clinical improvement AND absence of decrease of CRP level > 50%), 3 supplementary days of treatment at 400 mg/day will be done at D4, D5, D6 followed by a decrease at 200 mg/day at D7 and 100 mg/day at D8 and stop thereafter
Arm/Group | ANAKINRA -- Severe COVID Population (WHO-CPS =5) | Standard of Care -- Severe COVID Population (WHO-CPS =5) | ANAKINRA -- Critical COVID Population (WHO-CPS >5) | Standard of Care -- Critical COVID Population (WHO-CPS >5)
Number analyzed (Participants) | 59 | 55 | 22 | 20
percentage of participants
  Day 14 | 85 [76 to 94] | 76 [66 to 88] | 91 [80 to 100] | 85 [71 to 100]
  Day 28 | 78 [68 to 89] | 76 [66 to 88] | 96 [73 to 100] | 85 [71 to 100]
  Day 90 | 72 [61 to 85] | 72 [62 to 85] | 73 [56 to 94] | 80 [64 to 100]
Statistical Analysis 1: Comparison: ANAKINRA -- Severe COVID Population (WHO-CPS =5) vs Standard of Care -- Severe COVID Population (WHO-CPS =5); 14 days; Test type: Superiority; Regression, Cox; adjusted for age and centre; Hazard Ratio (HR) = 0.56, 95% CI 2-sided [0.23 to 1.29]
Statistical Analysis 2: Comparison: ANAKINRA -- Severe COVID Population (WHO-CPS =5) vs Standard of Care -- Severe COVID Population (WHO-CPS =5); 28 days; Test type: Superiority; Regression, Cox; Adjusted for age and centre; Hazard Ratio (HR) = 0.77, 95% CI 2-sided [0.33 to 1.77]
Statistical Analysis 3: Comparison: ANAKINRA -- Severe COVID Population (WHO-CPS =5) vs Standard of Care -- Severe COVID Population (WHO-CPS =5); Test type: Superiority — 90 days; Regression, Cox; adjusted on age and centre; Hazard Ratio (HR) = 0.97, 95% CI 2-sided [0.46 to 2.04] — % Confidence interval is % Credible interval here
Statistical Analysis 4: Comparison: ANAKINRA -- Critical COVID Population (WHO-CPS >5) vs Standard of Care -- Critical COVID Population (WHO-CPS >5); Test type: Superiority; Regression, Cox; adjusted on age and centre; Hazard Ratio (HR) = 0.64, 95% CI 2-sided [0.11 to 3.86]
Statistical Analysis 5: Comparison: ANAKINRA -- Critical COVID Population (WHO-CPS >5) vs Standard of Care -- Critical COVID Population (WHO-CPS >5); Test type: Superiority; Regression, Cox; adjusted on age and centre; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.19 to 4.68]
Statistical Analysis 6: Comparison: ANAKINRA -- Critical COVID Population (WHO-CPS >5) vs Standard of Care -- Critical COVID Population (WHO-CPS >5); Test type: Superiority; Regression, Cox; adjusted on age and centre; Cox Proportional Hazard = 1.22, 95% CI 2-sided [0.31 to 4.87]

7. Secondary Outcome: Mean of Ventilator Free-days at Day 28 -- Critical COVID Population (WHO-clinical Progression Scale >5 at Baseline)
Description: 28-day Ventilator Free-days
Time Frame: 28 days
Population: Critical COVID Population (WHO clinical progression scale >5 at baseline)
Measure: Mean (Standard Deviation); unit: days
Arm/Group | ANAKINRA -- Critical COVID Population (WHO-CPS >5) | Standard of Care -- Critical COVID Population (WHO-CPS >5)
Number analyzed (Participants) | 22 | 20
days | 14.4 (11.9) | 14.8 (12.6)
Statistical Analysis 1: Comparison: ANAKINRA -- Critical COVID Population (WHO-CPS >5) vs Standard of Care -- Critical COVID Population (WHO-CPS >5); Test type: Superiority; adjusted on age and centre; Mean Difference (Net) = -0.4, 95% CI 2-sided [-8.3 to 6.4]

8. Secondary Outcome: PaO2/FiO2 Ratio -- Critical COVID Population (WHO Clinical Progression Scale >5 at Baseline)
Description: Evolution of PaO2/FiO2 ratio
Time Frame: day 1 to day 14
Population: No statistical comparison was performed due to the limited number of patients with available follow-up data.
Measure: Median (Inter-Quartile Range); unit: mmHg
Arm/Group | ANAKINRA -- Critical COVID Population (WHO-CPS >5) | Standard of Care -- Critical COVID Population (WHO-CPS >5)
Number analyzed (Participants) | 11 | 10
mmHg
  Day 1 | 175.0 [117.9 to 225.0] | 118.7 [96.9 to 172.5]
  Day 4: number analyzed (Participants) | 10 | 8
  Day 4 | 114.5 [103.0 to 154.6] | 136.1 [98.1 to 282.1]
  Day 7: number analyzed (Participants) | 11 | 9
  Day 7 | 182.0 [163.0 to 262.6] | 142.0 [79.3 to 192.5]
  Day 14: number analyzed (Participants) | 5 | 6
  Day 14 | 180.0 [175.0 to 276.7] | 218.3 [139.4 to 272.5]

9. Secondary Outcome: Cumulative Incidence (Percentage of Participants) of Oxygen Supply Independency
Description: Time to oxygen supply independency
Time Frame: 28 and 90 days
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ANAKINRA -- Severe COVID Population (WHO-CPS =5) | Standard of Care -- Severe COVID Population (WHO-CPS =5) | ANAKINRA -- Critical COVID Population (WHO-CPS >5) | Standard of Care -- Critical COVID Population (WHO-CPS >5)
Number analyzed (Participants) | 59 | 55 | 22 | 20
percentage of participants
  Day 28 | 63 [49 to 74] | 69 [55 to 80] | 59 [35 to 77] | 50 [26 to 70]
  Day 90 | NA [NA to NA] — No assessment in Severe COVID Population (WHO Clinical Progression Scale =5 at baseline) at Day 90 | NA [NA to NA] — No assessment in Severe COVID Population (WHO Clinical Progression Scale =5 at baseline) at Day 90 | 77 [48 to 91] | 70 [43 to 86]
Statistical Analysis 1: Comparison: ANAKINRA -- Severe COVID Population (WHO-CPS =5) vs Standard of Care -- Severe COVID Population (WHO-CPS =5); Test type: Superiority; Fine-Gray model; Adjusted for age and centre; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.64 to 1.61]
Statistical Analysis 2: Comparison: ANAKINRA -- Critical COVID Population (WHO-CPS >5) vs Standard of Care -- Critical COVID Population (WHO-CPS >5); Test type: Superiority; Fine-Gray model — Adjusted for age and centre; Adjusted for age and centre; Hazard Ratio (HR) = 1.33, 95% CI 2-sided [0.58 to 3.07]

10. Secondary Outcome: Cumulative Incidence (Percentage of Participants) of Discharge From Hospital
Description: Time to discharge from hospital
Time Frame: 28 days
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ANAKINRA -- Severe COVID Population (WHO-CPS =5) | Standard of Care -- Severe COVID Population (WHO-CPS =5) | ANAKINRA -- Critical COVID Population (WHO-CPS >5) | Standard of Care -- Critical COVID Population (WHO-CPS >5)
Number analyzed (Participants) | 59 | 55 | 22 | 20
percentage of participants
  Day 28 | 58 [44 to 69] | 62 [47 to 73] | 41 [20 to 61] | 40 [18 to 61]
  Day 90 | NA [NA to NA] — No assessment in Severe COVID Population (WHO-CPS =5) at Day 90 | NA [NA to NA] — No assessment in Severe COVID Population (WHO-CPS =5) at Day 90 | 68 [42 to 84] | 65 [39 to 82]
Statistical Analysis 1: Comparison: ANAKINRA -- Severe COVID Population (WHO-CPS =5) vs Standard of Care -- Severe COVID Population (WHO-CPS =5); Test type: Superiority; Fine-Gray model; adjusted on age and centre; Hazard Ratio (HR) = 0.91, 95% CI 2-sided [0.56 to 1.48]
Statistical Analysis 2: Comparison: ANAKINRA -- Critical COVID Population (WHO-CPS >5) vs Standard of Care -- Critical COVID Population (WHO-CPS >5); Test type: Superiority; Fine-Gray model — adjusted on age and centre; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.35 to 2.34]

11. Secondary Outcome: Cumulative Incidence (Percentage of Participants) of Intensive Care Unit Discharge -- Critical COVID Population (WHO Clinical Progression Scale >5 at Baseline)
Description: Time to discharge from Intensive Care Unit
Time Frame: 28 and 90 days
Population: Patients in the intensive care unit at inclusion
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ANAKINRA -- Critical COVID Population (WHO-CPS >5) | Standard of Care -- Critical COVID Population (WHO-CPS >5)
Number analyzed (Participants) | 17 | 17
percentage of participants
  Day 28 | 65 [36 to 83] | 65 [36 to 93]
  Day 90 | 88 [47 to 98] | 82 [49 to 95]
Statistical Analysis 1: Comparison: ANAKINRA -- Critical COVID Population (WHO-CPS >5) vs Standard of Care -- Critical COVID Population (WHO-CPS >5); Day 28; Test type: Superiority; Fine-Gray model — adjusted on age and centre; Hazard Ratio (HR) = 1, 95% CI 2-sided [0.43 to 2.32]
Statistical Analysis 2: Comparison: ANAKINRA -- Critical COVID Population (WHO-CPS >5) vs Standard of Care -- Critical COVID Population (WHO-CPS >5); Day 90; Test type: Superiority; Fine-Gray model — adjusted on age and centre; Hazard Ratio (HR) = 1.09, 95% CI 2-sided [0.52 to 2.29]

ADVERSE EVENTS:
Time Frame: Adverse events were systematically assessed at Days 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13 and 14 while participants were inpatient, and at Days 28 and 60 and 90.
Description: Only deaths and serious adverse events were reported. "0" total Number of Participants at Risk means " Other (Not Including Serious) Adverse Events were not monitored/analyzed ".
Arm/Group | ANAKINRA -- Severe COVID Population (WHO-CPS =5) | Standard of Care -- Severe COVID Population (WHO-CPS =5) | ANAKINRA -- Critical COVID Population (WHO-CPS >5) | Standard of Care -- Critical COVID Population (WHO-CPS >5)
All-Cause Mortality (participants affected / at risk) | 16/59 | 16/55 | 6/22 | 4/20
Serious Adverse Events (participants affected / at risk) | 27/59 | 21/55 | 14/22 | 9/20
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ANAKINRA -- Severe COVID Population (WHO-CPS =5) (N=59) | Standard of Care -- Severe COVID Population (WHO-CPS =5) (N=55) | ANAKINRA -- Critical COVID Population (WHO-CPS >5) (N=22) | Standard of Care -- Critical COVID Population (WHO-CPS >5) (N=20)
Acute respiratory distress syndrom (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 12 (13) | 3 (3) | 4 (4)
Bacterial sepsis (Infections and infestations) | 7 (10) | 2 (4) | 6 (8) | 5 (10)
Hepatic cytolysis (Hepatobiliary disorders) | 7 (7) | 0 (0) | 0 (0) | 0 (0)
Multiple organ failure (General disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Vascular disorders) | 2 (3) | 1 (1) | 1 (1) | 0 (0)
Acute renal failure (Renal and urinary disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 3 (3) | 0 (0)
Coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholestatis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fungal sepsis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Myelomia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sudden death (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Arterial ischaemia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thombopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Complication of intubation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metastatic progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Herpetic pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Olgivie syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Undertermined sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabete (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Meningo-radiculitus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Heart failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-14): https://cdn.clinicaltrials.gov/large-docs/84/NCT04341584/Prot_SAP_001.pdf